CLINICAL TRIAL: NCT05932160
Title: Research Investigator
Brief Title: Effect of Intravenous Dextrose on PONV in Patients Undergoing Gynecological Laparoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weifang Medical University (Other)
Responsible Party: Principal Investigator, Jiang Liu, Research investigator, Weifang Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023YX104
Record Dates: First submitted 2023-06-06; First posted 2023-07-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Glucose; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Patients in the experimental group were infused intravenously with 5% dextrose (400 ml/h) in the PACU. The study outcomes were collected at three assessment periods, 0-0.5 h, 0.5-6 h, 6-24 h, after anesthesia by an independent investigator.
  Interventions: Other: 5% glucose
- Control group (Active Comparator): Patients in the control group were infused intravenously with ringer lactate solution (400 ml/h) in the PACU. The study outcomes were collected at three assessment periods, 0-0.5 h, 0.5-6 h, 6-24 h, after anesthesia by an independent investigator.
  Interventions: Other: lactated ringers

INTERVENTIONS:
Other: 5% glucose — Patients in the experimental group were infused intravenously with 5% dextrose (500 ml/h) in the PACU.
  Other Names: 5% dextrose
  Arms: Experimental group
Other: lactated ringers — Patients in the control group were infused intravenously with lactated ringers (500 ml/h) in the PACU.
  Arms: Control group

SUMMARY:
This study is to explore the relationship between intravenous infusion of dextrose during emergence from anesthesia and the incidence of PONV in patients undergoing gynecology laparoscopy (GL).

ELIGIBILITY:
Inclusion Criteria:

1. ASA I or II;
2. Performing gynecologic laparoscopic procedures under general anesthesia;

Exclusion Criteria:

1. age <18 or >75
2. severe hypertension,diabetes mellitus, significant hepatic or renal disease
3. inability to follow protocol
4. refusal to participant

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | Measured at 0.5 hours postoperatively.
  The severity and incidence of PONV at 0.5 hours postoperatively.
Postoperative nausea and vomiting | Measured at 2 hours postoperatively.
  The severity and incidence of PONV at 2 hours postoperatively.
Postoperative nausea and vomiting | Measured at 24 hours postoperatively.
  The severity and incidence of PONV at 24 hours postoperatively.

SECONDARY OUTCOMES:
Consumption of postoperative analgesic | Approximately 24 hours after surgery.
  Record the type and dosage of postoperative analgesic within 24 hours after surgery.
Postoperative pain response | Measured at 0.5 hours postoperatively.
  The Visual Analog Score was used to assess pain response at 0.5 hours postoperatively.
  The score ranges from 0 (pain free or no pain) to 10 (worst pain).
Postoperative pain response | Measured at 2 hours postoperatively.
  The Visual Analog Score was used to assess pain response at 2 hours postoperatively.
  The score ranges from 0 (pain free or no pain) to 10 (worst pain).
Postoperative pain response | Measured at 24 hours postoperatively.
  The Visual Analog Score was used to assess pain response at 24 hours postoperatively.
  The score ranges from 0 (pain free or no pain) to 10 (worst pain).
Recovery time of PACU | Approximately 24 hours after surgery.
  Record PACU recovery time in hours. The criteria for discharge from PACU was the achievement of a modified Aldrete score ≥ 9.
Consumption of postoperative rescue antiemetic | Approximately 24 hours after surgery.
  Record the type and dosage of postoperative rescue antiemetic within 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Liu, B.S, Principal Investigator — Weifang Medical University
Locations (1):
- Jiang Liu, Weifang, Shandong, China

IPD SHARING:
Plan to Share IPD: No